CLINICAL TRIAL: NCT00005696
Title: Early Atherosclerosis Change in Two Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4263; R01HL049885 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2005-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Carotid Artery Diseases; Coronary Disease; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Carotid Artery Diseases; Coronary Disease; Atherosclerosis

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To complete end point analysis for the Monitored Atherosclerosis Regression Study (MARS) and to compare coronary versus carotid treatment effect relationships in MARS to coronary versus carotid treatment effect relationships in the Cholesterol Lowering Atherosclerosis Study (CLAS). Both MARS and CLAS were serial arterial imaging trials that explored the reversibility of atherosclerosis with lipid-lowering therapy in native coronary, carotid, and femoral arterial beds, as well as in coronary artery bypass grafts.

DETAILED DESCRIPTION:
BACKGROUND:

MARS was a randomized, double-blind, placebo-controlled, angiographic trial comparing the effects of lipid lowering by lovastatin and diet with diet plus placebo in 270 subjects. The target study population consisted of males and females under 70 years of age with cholesterol levels from 200 to 295 mg/dL and coronary artery disease in two or more coronary artery segments. Follow-up coronary angiograms were performed two and four years post-randomization in 247 and 68 subjects, respectively; providing information on atherosclerosis regression/progression of coronary artery intrusive lesions. Carotid ultrasound images have been recorded at four month intervals for periods up to four years in 215 subjects providing information on atherosclerosis regression/progression of pre-intrusive (intima-media thickness) lesions in parallel with coronary artery intrusive lesions. Unique features of MARS included: 1) Simultaneous coronary angiography (evaluated both by quantitative coronary angiography (QCA) and panel-reading) and carotid ultrasonography in a cohort of over 200 subjects; 2) The opportunity to evaluate the largest lipoprotein and apolipoprotein data collected in an angiographic trial to date. This included extensive VLDL, LDL, IDL, and HDL subclasses as well as LDL type pattern, lipoprotein particles and apolipoprotein (including AI, B, CIII, and E); and, 3) The opportunity to evaluate dietary effects on atherosclerosis regression/progression only in one other angiographic trail, CLAS.

The Cholesterol Lowering Atherosclerosis Study (CLAS) was a randomized angiographic trial comparing combined colestipol/niacin therapy with placebo in 162 subjects. A unique feature of MARS and CLAS has shown a similar effect in CLAS-like men (non-smoking men with CABG) and women. Since carotid intima-media thickness, QCA, and global change score have been shown to be predictive of clinical coronary events, understanding the relationship between these atherosclerotic measures may be important in establishing carotid intima-media thickness measurements as a proxy measure for coronary atherosclerosis.

DESIGN NARRATIVE:

Collected data for both trials were analyzed and compared to evaluate effects of treatment on carotid and coronary artery atherosclerotic lesions. Coronary angiograms and carotid ultrasound imaging were performed under identical conditions in both trials. Five major databases were available for analysis, including: the coronary artery database (QCA processed); the carotid artery database (ultrasound evaluation); the coronary artery database (panel evaluation); the nutrient content database, and the clinical and biochemical database. Major comparisons included measurements of atherosclerotic lesions in both arteries, the effects of lipid, lipoprotein, and apolipoprotein levels on vascular lesions, and the effect of nutrient intake (in particular total fat, saturated fat, and cholesterol) on rates of measured lesion change. Additional associations were sought between preintrusive carotid lesions and intrusive coronary lesions between males and females, smokers and nonsmokers, differences in age, and differential drug effect on HDL-cholesterol.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-01; Study Completion 1996-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hodis — University of Southern California

REFERENCES:
- [Background] Alaupovic P, Mack WJ, Knight-Gibson C, Hodis HN. The role of triglyceride-rich lipoprotein families in the progression of atherosclerotic lesions as determined by sequential coronary angiography from a controlled clinical trial. Arterioscler Thromb Vasc Biol. 1997 Apr;17(4):715-22. doi: 10.1161/01.atv.17.4.715. PMID 9108785
- [Background] Alaupovic P, Hodis HN, Knight-Gibson C, Mack WJ, LaBree L, Cashin-Hemphill L, Corder CN, Kramsch DM, Blankenhorn DH. Effects of lovastatin on ApoA- and ApoB-containing lipoproteins. Families in a subpopulation of patients participating in the Monitored Atherosclerosis Regression Study (MARS). Arterioscler Thromb. 1994 Dec;14(12):1906-13. doi: 10.1161/01.atv.14.12.1906. PMID 7981178
- [Background] Hodis HN, Mack WJ, Dunn M, Liu C, Liu C, Selzer RH, Krauss RM. Intermediate-density lipoproteins and progression of carotid arterial wall intima-media thickness. Circulation. 1997 Apr 15;95(8):2022-6. doi: 10.1161/01.cir.95.8.2022. PMID 9133510
- [Background] Markus RA, Mack WJ, Azen SP, Hodis HN. Influence of lifestyle modification on atherosclerotic progression determined by ultrasonographic change in the common carotid intima-media thickness. Am J Clin Nutr. 1997 Apr;65(4):1000-4. doi: 10.1093/ajcn/65.4.1000. PMID 9094885
- [Background] Hodis HN. Reversibility of atherosclerosis--evolving perspectives from two arterial imaging clinical trials: the cholesterol lowering atherosclerosis regression study and the monitored atherosclerosis regression study. J Cardiovasc Pharmacol. 1995;25 Suppl 4:S25-31. PMID 8907211
- [Background] Mack WJ, Hodis HN. Efficacy of interventions designed to inhibit the progression of coronary atherosclerosis. Diabetes Res Clin Pract. 1996 Feb;30 Suppl:37-53. doi: 10.1016/s0168-8227(96)80037-4. PMID 8964192
- [Background] Mack WJ, Krauss RM, Hodis HN. Lipoprotein subclasses in the Monitored Atherosclerosis Regression Study (MARS). Treatment effects and relation to coronary angiographic progression. Arterioscler Thromb Vasc Biol. 1996 May;16(5):697-704. doi: 10.1161/01.atv.16.5.697. PMID 8963728
- [Background] Hodis HN, Mack WJ, LaBree L, Selzer RH, Liu C, Liu C, Alaupovic P, Kwong-Fu H, Azen SP. Reduction in carotid arterial wall thickness using lovastatin and dietary therapy: a randomized controlled clinical trial. Ann Intern Med. 1996 Mar 15;124(6):548-56. doi: 10.7326/0003-4819-124-6-199603150-00002. PMID 8597317
- [Background] Shircore AM, Mack WJ, Selzer RH, Lee PL, Azen SP, Alaupovic P, Hodis HN. Compensatory vascular changes of remote coronary segments in response to lesion progression as observed by sequential angiography from a controlled clinical trial. Circulation. 1995 Nov 1;92(9):2411-8. doi: 10.1161/01.cir.92.9.2411. PMID 7586339
- [Background] Hodis HN, Mack WJ. Triglyceride-rich lipoproteins and the progression of coronary artery disease. Curr Opin Lipidol. 1995 Aug;6(4):209-14. doi: 10.1097/00041433-199508000-00004. PMID 7670749
- [Background] Hodis HN, Mack WJ, LaBree L, Cashin-Hemphill L, Sevanian A, Johnson R, Azen SP. Serial coronary angiographic evidence that antioxidant vitamin intake reduces progression of coronary artery atherosclerosis. JAMA. 1995 Jun 21;273(23):1849-54. PMID 7776501
- [Background] Hodis HN, Mack WJ, Azen SP, Alaupovic P, Pogoda JM, LaBree L, Hemphill LC, Kramsch DM, Blankenhorn DH. Triglyceride- and cholesterol-rich lipoproteins have a differential effect on mild/moderate and severe lesion progression as assessed by quantitative coronary angiography in a controlled trial of lovastatin. Circulation. 1994 Jul;90(1):42-9. doi: 10.1161/01.cir.90.1.42. PMID 8026027
- [Background] Mack WJ, Azen SP, Dunn M, Hodis HN. A comparison of quantitative computerized and human panel coronary endpoint measures: implications for the design of angiographic trials. Control Clin Trials. 1997 Apr;18(2):168-79. doi: 10.1016/s0197-2456(96)00181-x. PMID 9129860
- [Background] Azen SP, Qian D, Mack WJ, Sevanian A, Selzer RH, Liu CR, Liu CH, Hodis HN. Effect of supplementary antioxidant vitamin intake on carotid arterial wall intima-media thickness in a controlled clinical trial of cholesterol lowering. Circulation. 1996 Nov 15;94(10):2369-72. doi: 10.1161/01.cir.94.10.2369. PMID 8921775
- [Background] Azen SP, Mack WJ, Cashin-Hemphill L, LaBree L, Shircore AM, Selzer RH, Blankenhorn DH, Hodis HN. Progression of coronary artery disease predicts clinical coronary events. Long-term follow-up from the Cholesterol Lowering Atherosclerosis Study. Circulation. 1996 Jan 1;93(1):34-41. doi: 10.1161/01.cir.93.1.34. PMID 8616937
- [Background] Vigen C, Hodis HN, Selzer RH, Mahrer PR, Mack WJ. Relation of progression of coronary artery atherosclerosis to risk of cardiovascular events (from the Monitored Atherosclerosis Regression Study). Am J Cardiol. 2005 Jun 1;95(11):1277-82. doi: 10.1016/j.amjcard.2005.01.068. PMID 15904629